CLINICAL TRIAL: NCT03815461
Title: Phase II Clinical Study of Nab-paclitaxel Combined With S-1 as Induction Therapy for Locally Advanced Pancreatic Cancer
Brief Title: Nab-paclitaxel Combined With S-1 as Induction Therapy for Locally Advanced Pancreatic Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Chinese Academy of Medical Sciences (Other)
Responsible Party: Principal Investigator, Aiping Zhou, Cancer Hospital & Institute, Chinese Academy of Medical Sciences
Organization: ChineseAMS (Unknown)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CSPC-KAL-PC-05
Record Dates: First submitted 2019-01-23; First posted 2019-01-24 (Actual); Last update posted 2019-01-25 (Actual); Status verified 2019-01

CONDITIONS: Locally Advanced Pancreatic Cancer
MeSH Terms: interventions — 130-nm albumin-bound paclitaxel; S 1 (combination)

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- experiment group (Experimental): Nab-paclitaxel+S-1
  Interventions: Drug: Nab-paclitaxel and S-1

INTERVENTIONS:
Drug: Nab-paclitaxel and S-1 — Nab-paclitaxel was administered at 125mg/m2 intravenously on day 1 and 8, S-1 （80, 100, or 120 mg/d according to body-surface area on days 1 through 14 of a 21-day cycle for 4-6 cycles.

SUMMARY:
This single-arm, Phase II clinical trial is to evaluate the efficacy and safety of nab-paclitaxel plus S-1 in locally advanced pancreatic cancer who were borderline resectable or unresectable .

DETAILED DESCRIPTION:
This single-arm, Phase II clinical trial is to evaluate the efficacy and safety of nab-paclitaxel plus S-1 in locally advanced pancreatic cancer who were borderline resectable or unresectable . Nab-paclitaxel was administered at 125mg/m2 intravenously on day 1 and 8, S-1 （80, 100, or 120 mg/d according to body-surface area on days 1 through 14 of a 21-day cycle for 4-6 cycles.

During the study, if the subject's weight change was ≤10% from baseline, the dose was calculated based on the measured value at baseline. If the change was >10%, the body surface area of the subject should be recalculated and the dose administered should be adjusted. .

Study treatment period Borderline resectable: According to the results of imaging examination, MDT discussed to determine the surgical resectability and timing of surgery. The chemotherapy time was 4-6 cycles.

Unresectable: Chemotherapy for up to 6 cycles. According to the results of imaging examination, MDT determined the resectability of the operation. It was decided by the investigator and the patient to continue chemotherapy (S-1 maintenance), surgery or radiotherapy.

ELIGIBILITY:
Inclusion Criteria:

* patient compliance is good, the research process of this study can be understood, and written informed consent is signed;
* Age ≥ 18 years old, ≤ 75 years old;
* Histologically or cytologically confirmed pancreatic adenocarcinoma；
* no prior treatment;
* Based on imaging findings, MDT decided patients intoborderline resectable (group A) or unresectable (group B) (according to the resectability assessment criteria in the 2018 Pancreatic Cancer Comprehensive Care Guidelines);
* ECOG<2;
* Bone marrow function: hemoglobin (HGB) ≥ 90g / L; absolute neutrophil count (ANC) ≥ 1.5 × 109 / L; platelets (PLT) ≥ 100 × 109 / L;
* Liver function: ALT, AST ≤ 2.5 × upper limit of normal (ULN), if there is liver metastasis, ALT, AST ≤ 5 × ULN; serum total bilirubin < 1.5 × ULN;
* Renal function: serum creatinine is within normal range;
* Patients without biliary obstruction, patients requiring biliary stent implantation must be completed at least 7 days prior to enrollment;
* Non-pregnant and lactating women, women of reproductive age/male should take effective contraceptive measures during the study period and within 6 months after the end of the study treatment;
* No contraindication to the use of S-1and albumin-bound paclitaxel.

Exclusion Criteria:

* Patients who have had other malignant tumors within 5 years (except for cured cervical cancer in situ or non-melanoma skin cancer);
* Interstitial pneumonia or pulmonary fibrosis;
* Severe pleural effusion or ascites;
* Watery diarrhea;
* There are serious concomitant diseases: such as HIV-positive,chronic HBV/HCV in active period, people who have diabetes and poorly controlled by hypoglycemic drugs, clinically severe (ie, active) heart disease, uncontrolled epilepsy, central nervous system disease or mental disorder;
* Current or previous patients with grade II peripheral neuropathy;
* Abnormal digestive tract or metabolic function, which may affect the s-1 absorber;
* Participated in other clinical researchers within 4 weeks prior to enrollment;
* Patients who have undergone organ transplantation;
* Patients considered by the investigator to be unfit for this trial.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2019-02-01 (Estimated); Primary Completion 2023-06-01 (Estimated); Study Completion 2023-10-02 (Estimated)

PRIMARY OUTCOMES:
PFS | up to 2.5 years

SECONDARY OUTCOMES:
R0 resection rate | 6 months
Overall survival rate | 2 years
Overall survival | up to 2.5 years
Adverse reaction rate | up to 2.5 years

CONTACTS AND LOCATIONS:
Overall Officials: Zhou Aiping, Principal Investigator — National Cancer Center/Cancer Hospital, China
Locations (1):
- National Cancer Center/Cancer Hospital, Chinese Academy of Medical Sciences and Peking Union Medical College, Beijing, China